CLINICAL TRIAL: NCT03527459
Title: Implementing an Interpersonal Theory of Suicide Treatment Approach to Improve Outcomes in Suicidal Youth
Brief Title: Implementing an IPTS Treatment Approach to Improve Outcomes in Suicidal Youth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Sunita Stewart, Professor, University of Texas Southwestern Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GA2016-010
Record Dates: First submitted 2018-05-02; First posted 2018-05-17 (Actual); Last update posted 2019-11-01 (Actual); Status verified 2019-10

CONDITIONS: Suicidal Ideation; Depression
MeSH Terms: conditions — Suicidal Ideation; Depression

STUDY DESIGN:
Intervention Model Description: Half of the clients in the SPARC clinical program are enrolled into either the original program or SPARC B (which will overlap significantly with SPARC A but targets in some sessions specific negative cognitions of perceived burdensomeness). The program is already structured so that each patient consistently attends either a morning or an afternoon track, with different therapists running each track. This allows for separate programs in each track. Clinically justifiable innovations are routinely introduced into the program usually in a stepwise fashion in one or another part by one set of therapists at a time. We will assess relative impact of SPARC A and SPARC B on depressive symptoms and suicide ideation. Our investigation will allow us to assess whether this innovation is effective. Patients will not be randomized at the individual level, but rather their time slot (usually decided based on opening within the program) will place them into either SPARC A or SPARC B.
Who Masked: Participant, Care Provider
Masking Description: Participants are masked as to the treatment arm to which they are assigned. Care providers in the control arm are masked to the interventions being tested in the experimental arm, so as to not inadvertently deliver aspects of SPARC B intervention to the SPARC A group. The outcomes assessor is not collecting primary outcome data, which is self-reported via online survey.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SPARC A (Active Comparator): SPARC A is an existing clinical program which has a general focus on negative cognitions.
  Interventions: Behavioral: SPARC A
- SPARC B (Experimental): SPARC B includes all aspects of the SPARC A clinical program, but targets negative cognitions of perceived burdensomeness in some sessions.
  Interventions: Behavioral: SPARC B

INTERVENTIONS:
Behavioral: SPARC B — SPARC B includes all aspects of the SPARC A clinical program, as well as targeting negative cognitions of perceived burdensomeness.
  Arms: SPARC B
Behavioral: SPARC A — SPARC A is an existing clinical program with a general focus on negative cognitions.
  Arms: SPARC A

SUMMARY:
The purpose of this project is to evaluate a set of interventions derived from a theory of suicide that supplements a clinical program and compare their effects on outcomes to the outcomes of the unsupplemented program. This study proposes to evaluate the effect of these interventions on reducing specific negative cognitions associated with depression and suicide ideation in an intensive outpatient program for suicidal youth (Suicide Prevention and Resilience at Children's, SPARC).

DETAILED DESCRIPTION:
The trial will be conducted in a program where half of the clients are enrolled into either the original program (SPARC A which has a general focus on negative cognitions) or SPARC B (which will overlap significantly with SPARC A but targets in some sessions specific negative cognitions of perceived burdensomeness). The program is already structured so that each patient consistently attends either a morning or an afternoon track, with different therapists running each track. This allows for separate programs in each track. Clinically justifiable innovations are routinely introduced into the program usually in a stepwise fashion in one or another part by one set of therapists at a time. The investigators propose to take advantage of this partial introduction by assessing relative impact of SPARC A and SPARC B on depressive symptoms and suicide ideation. The investigators have no data to indicate that one program will be better than the other. The investigation will, however, allow the investigators to assess whether this innovation in fact is effective. Patients will not be randomized at the individual level, but rather their time slot (usually decided based on opening within the program) will place them into either SPARC A or SPARC B. The two programs are of identical length with numerous features in common, differing only in the specificity of the exercises and examples and their relevance to perceived burdensomeness. Routine assessments at entry and discharge from the program will not change based on study enrollment. However, suicide ideation, depressive symptoms, and negative cognitions (perceived burdensomeness and thwarted belongingness) will be more formally assessed at the one-month follow-up meeting or phone call which will add approximately 10 minutes to the contact.

ELIGIBILITY:
Inclusion Criteria:

* adolescents, ages 12 - 17
* enrolled in the SPARC program at Children's Medical Center of Dallas
* completed at least 5 SPARC group therapy sessions

Exclusion Criteria:

* adolescents who have previously received treatment in the control arm of the study

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 123 (Actual)
Dates: Start 2017-11-14 (Actual); Primary Completion 2019-03-07 (Actual); Study Completion 2019-06-01 (Actual)

PRIMARY OUTCOMES:
Interpersonal Needs Questionnaire (INQ) (Van Orden et al., 2012) | through program completion, an average of 6 weeks
  change in perceived burdensomeness
Concise Health Risk Tracking Self Report (CHRT-SR) (Trivedi et al., 2011) | through program completion, an average of 6 weeks
  suicide ideation (self-report)

SECONDARY OUTCOMES:
Quick Inventory of Depressive Symptomatology - Adolescent Version Self-Report (QIDS-A-SR-16) (Bernstein et al., 2010) | through program completion, an average of 6 weeks
  change in depressive symptoms
Interpersonal Needs Questionnaire (INQ) (Van Orden et al., 2012) | 1 month after program completion
  change in perceived burdensomeness
Concise Health Risk Tracking Self Report (CHRT-SR) (Trivedi et al., 2011) | 1 month after program completion
  change in suicide ideation (self-report)
Quick Inventory of Depressive Symptomatology - Adolescent Version Self-Report (QIDS-A-SR-16) (Bernstein et al., 2010) | 1 month after program completion
  change in depressive symptoms
Concise Health Risk Tracking Self Report (CHRT-SR) | between program completion, an average of 6 weeks, and 1 month after program completion
  change in suicide ideation (self-report)

CONTACTS AND LOCATIONS:
Overall Officials: Sunita M. Stewart, PhD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- Children's Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bernstein IH, Rush AJ, Trivedi MH, Hughes CW, Macleod L, Witte BP, Jain S, Mayes TL, Emslie GJ. Psychometric properties of the Quick Inventory of Depressive Symptomatology in adolescents. Int J Methods Psychiatr Res. 2010 Dec;19(4):185-94. doi: 10.1002/mpr.321. PMID 20683845
- [Background] Trivedi MH, Wisniewski SR, Morris DW, Fava M, Gollan JK, Warden D, Nierenberg AA, Gaynes BN, Husain MM, Luther JF, Zisook S, Rush AJ. Concise Health Risk Tracking scale: a brief self-report and clinician rating of suicidal risk. J Clin Psychiatry. 2011 Jun;72(6):757-64. doi: 10.4088/JCP.11m06837. PMID 21733476
- [Background] Van Orden KA, Cukrowicz KC, Witte TK, Joiner TE. Thwarted belongingness and perceived burdensomeness: construct validity and psychometric properties of the Interpersonal Needs Questionnaire. Psychol Assess. 2012 Mar;24(1):197-215. doi: 10.1037/a0025358. Epub 2011 Sep 19. PMID 21928908